CLINICAL TRIAL: NCT05830214
Title: Digital Smartwatch Measurements as Potential Biomarkers for Remote Disease Tracking in ALS (CAPTURE ALS Smarwatch)
Brief Title: Digital Smartwatch Measurements as Potential Biomarkers for Remote Disease Tracking in ALS
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty procuring study device
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00125737
Record Dates: First submitted 2023-02-24; First posted 2023-04-26 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Muscular Atrophy, Progressive; Frontotemporal Dementia; Healthy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Muscular Atrophy, Spinal; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will use new smartwatch technology to continuously and remotely monitor the health of ALS patients and healthy controls over time. This information will be used to develop digital biomarkers for ALS.

DETAILED DESCRIPTION:
This is an optional study that is conducted in parallel to CAPTURE ALS (NCT05204017). In this exploratory, prospective, longitudinal study, CAPTURE ALS participants undergo remote physiological data collection using smartwatch technology. Participants will wear a specialized smartwatch (Health Gauge AI-Based Wearable Device ) for the duration of the study. ALS patients will be followed for 12 months, healthy controls will be followed for 8 months. Digital questionnaires will monitor participant-related outcomes bi-monthly. Gait assessments will be performed by ambulatory patients and healthy controls in clinic during CAPTURE ALS study visits to measure changes in walking activity.

ELIGIBILITY:
[PATIENTS]

Inclusion Criteria:

* Has ALS, classified as definite, probable, laboratory-supported probable, or possible ALS according to the revised El Escorial criteria or a related neurodegenerative disorder including ALS-FTD, PLS, PMA or asymptomatic individuals with a known ALS mutation (as previously confirmed during the individual's regular clinical care)
* Is the age of majority in their province of residence/treatment
* Has the cognitive capacity to provide informed consent
* Has proficiency in English or French in order to understand study instructions and respond to questionnaires

Exclusion Criteria:

* Is pregnant
* Has a history of active (clinically significant) skin disorders
* Has a history of allergic response to plastic materials
* Has an electronic implant of any kind (e.g. pacemaker)
* Has broken, damaged or irritated skin or rashes near the sensor application sites
* Is unstably housed or lack reliable contact information.
* Investigator judges that device retrieval will be difficult or unlikely
* Does not have a smartphone that will support the HG application
* Does not have daily access to a wireless connection

[HEALTHY CONTROLS]

Inclusion Criteria:

* Be between the ages of 40-80 unless age matched to a patient (+/-3 years) who is already enrolled.
* Is the age of majority in their province of residence/treatment
* Has the cognitive capacity to provide informed consent
* Has proficiency in English or French in order to understand study instructions and respond to questionnaires

Exclusion Criteria:

* Has a history of a neurological disease, including Central Nervous System disease (e.g., stroke, head injury, epilepsy) or Peripheral Nervous System disease (neuropathy, myopathy).
* Has a history of psychiatric disease (e.g., depression, bipolar disease) that is clinically diagnosed and/or with the current use of psychiatric medications (e.g., antidepressants) for an indication of a psychiatric disease.
* Is pregnant
* Has a history of active (clinically significant) skin disorders
* Has a history of allergic response to plastic materials
* Has an electronic implant of any kind (e.g. pacemaker)
* Has broken, damaged or irritated skin or rashes near the sensor application sites
* Is unstably housed or lack reliable contact information.
* Investigator judges that device retrieval will be difficult or unlikely
* Does not have a smartphone that will support the HG application
* Does not have daily access to a wireless connection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People living with ALS and related motor neuron diseases including ALS-Frontotemporal Dementia (ALS-FTD), Primary Lateral Sclerosis (PLS), Progressive Muscular Atrophy (PMA) and asymptomatic individuals with a known ALS mutation
  AND
  Healthy controls that are age and sex matched to patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Body Temperature | Up to 1 year
  Body temperature in Degrees Celsius as measured by the Health Gauge smartwatch worn by the participant
Respiratory rate | Up to 1 year
  Respiratory rate in breaths per minute as measured by the Health Gauge smartwatch worn by the participant
Oxygen saturation | Up to 1 year
  Oxygen saturation in percent as measured using the Health Gauge smartwatch worn by participants
Heart rate | Up to 1 year
  Heart rate in beats per minute as measured using the Health Gauge smartwatch worn by participants
Step count | Up to 1 year
  Physical activity in step count as measured using the Health Gauge smartwatch worn by participants
Distance travelled | Up to 1 year
  Physical activity in distance travelled (meters) as measured using the Health Gauge smartwatch worn by participants
Calories | Up to 1 year
  Physical activity in calories as measured using the Health Gauge smartwatch worn by participants
Sleep stage | Up to 1 year
  Sleep stage in time in wake, light and deep stages as measured using the Health Gauge smartwatch worn by participants

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | Baseline
  The TUG is used to assess changes in functional mobility. Participants arise from a chair, walk forward 3 meters, turn around, walk back to the chair and sit. The time to complete the test is measured.
Timed Up and Go (TUG) | Month 4
  The TUG is used to assess changes in functional mobility. Participants arise from a chair, walk forward 3 meters, turn around, walk back to the chair and sit. The time to complete the test is measured.
Timed Up and Go (TUG) | Month 8
  The TUG is used to assess changes in functional mobility. Participants arise from a chair, walk forward 3 meters, turn around, walk back to the chair and sit. The time to complete the test is measured.
Timed Up and Go (TUG) | Month 12
  The TUG is used to assess changes in functional mobility. Participants arise from a chair, walk forward 3 meters, turn around, walk back to the chair and sit. The time to complete the test is measured.
10 Meter Walk | Baseline
  The 10 Meter Walk Test is a performance measure used to assess walking speed over a short distance. This task will be performed with and without serial 3s subtraction. The time to walk 10 meters and the number of errors in the mental task are measured.
10 Meter Walk | 4 Months
  The 10 Meter Walk Test is a performance measure used to assess walking speed over a short distance. This task will be performed with and without serial 3s subtraction. The time to walk 10 meters and the number of errors in the mental task are measured.
10 Meter Walk | 8 Months
  The 10 Meter Walk Test is a performance measure used to assess walking speed over a short distance. This task will be performed with and without serial 3s subtraction. The time to walk 10 meters and the number of errors in the mental task are measured.
10 Meter Walk | 12 Months
  The 10 Meter Walk Test is a performance measure used to assess walking speed over a short distance. This task will be performed with and without serial 3s subtraction. The time to walk 10 meters and the number of errors in the mental task are measured.
2-Minute Timed Walk Test (2MWT) | Baseline
  The 2MWT assess overall gait function and endurance. The total distance travelled in 2 minutes is measured.
2-Minute Timed Walk Test (2MWT) | 4 Months
  The 2MWT assess overall gait function and endurance. The total distance travelled in 2 minutes is measured.
2-Minute Timed Walk Test (2MWT) | 8 Months
  The 2MWT assess overall gait function and endurance. The total distance travelled in 2 minutes is measured.
2-Minute Timed Walk Test (2MWT) | 12 Months
  The 2MWT assess overall gait function and endurance. The total distance travelled in 2 minutes is measured.
Changes in ALS Assessment Questionnaire (ALSAQ-40) Mobility Sub-score | Changes from baseline at 1 year
  Changes in self-reported physical mobility over 1 year as measured using the ALSAQ-40 mobility sub-score, lower scores indicate better mobility.
Changes in Generalized Anxiety Disorder 7 (GAD-7) score | Changes from baseline at 1 year
  Changes in self-reported anxiety over 1 year as measured using the GAD-7. The total score for the 7 items ranges from 0-21, with 0-4 (none to minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), 15-21 (severe anxiety).
Changes in ALSFRS-R Dyspnea and Orthopnea sub-scores | Changes from baseline at 1 year
  Changes in self-reported dyspnea and orthopnea over 1 year as measured using the ALS Functional Rating Scale dyspnea and orthopnea sub-scores. Each question is scored by the participant as "4" (never) to "0" (all of the time).
Changes in Patient Health Questionnaire (PHQ-9) score | Changes from baseline at 1 year
  Changes in self-reported depression over 1 year as measured using the PHQ-9. The total score for the 9 items ranges from 0-27, with 0-4 (none-minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), 20-27 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Jake Hayward, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada